CLINICAL TRIAL: NCT06153602
Title: Effectiveness of Intrathecal Nalbuphine as an Adjuvant to Subarachnoid Block on Postoperative Analgesia in Patients Undergoing Transurethral Resection of the Prostate
Brief Title: Effectiveness of Nalbuphine as an Adjuvant to Subarachnoid Block on Postoperative Analgesia in TURP Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 703/66
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2023-11

CONDITIONS: Transurethral Resection of Prostate
Keywords: Anesthesia, Spinal; Pain, Postoperative; Nalbuphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Nalbuphine; Sodium Chloride; Injections; Bupivacaine; Acetaminophen; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nalbuphine group (Experimental): 0.5% Hyperbaric or Isobaric Spinal Bupivacaine 5-20 mg (1-4 ml) + Nalbuphine(10mg/ml) 0.8 mg intrathecal
  Interventions: Drug: Nalbuphine Hydrochloride 10 MG/ML; Drug: Bupivacaine Hydrochloride, Spinal; Drug: Nalbuphine Hcl 10Mg/Ml Inj; Drug: Acetaminophen 500Mg Tab; Drug: Ondansetron 8mg
- Control group (Placebo Comparator): 0.5% Hyperbaric or Isobaric Spinal Bupivacaine 5-20 mg (1-4 ml) + 0.9% Sodium chloride 0.08 ml intrathecal
  Interventions: Drug: Sodium Chloride 0.9 % in 5 ML Injection; Drug: Bupivacaine Hydrochloride, Spinal; Drug: Nalbuphine Hcl 10Mg/Ml Inj; Drug: Acetaminophen 500Mg Tab; Drug: Ondansetron 8mg

INTERVENTIONS:
Drug: Nalbuphine Hydrochloride 10 MG/ML — Nalbuphine(10mg/ml) 0.8 mg intrathecal
  Arms: Nalbuphine group
Drug: Sodium Chloride 0.9 % in 5 ML Injection — 0.9% Sodium Chloride 0.08 ml intrathecal
  Arms: Control group
Drug: Bupivacaine Hydrochloride, Spinal — 0.5% Hyperbaric or Isobaric Spinal Bupivacaine 1-4 ml intrathecal
Drug: Nalbuphine Hcl 10Mg/Ml Inj — 4 mg IV prn for postoperative pain score>=4 q 6 h
Drug: Acetaminophen 500Mg Tab — 1 tab oral prn for postoperative pain score 1-3 q 6 h
Drug: Ondansetron 8mg — 8 mg IV prn for nausea or vomiting q 8 h

SUMMARY:
The goal of this clinical trial is to compare pain after surgery in patients undergoing Transurethral Resection of Prostate. The main question it aims to answer are: Intrathecal nalbuphine as an adjuvant to local anesthetic will better provide pain relief after TURP surgery.

Participants will be given a combination of nalbuphine and local anesthetic when getting a spinal block. Researchers will compare control group, given look-alike solution that contains no active drug to see if nalbuphine will better provide pain relief after surgery.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and side effects of nalbuphine, with the goal of providing anesthesiologists with evidence-based guidance for selecting the most appropriate pharmacological agents for their patients.

Participants will be given a combination of nalbuphine and local anesthetic when getting a spinal block. Researchers will compare control group, given look-alike solution that contains no active drug to see if nalbuphine will better provide pain relief after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for Transurethral Resection of Prostate under spinal anesthesia
* American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Allergy to study medications or hypersensitive to local anesthetics
* Contraindicated for neuraxial anesthesia
* Inability to self-report pain
* Chronic opioid used

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
VAS Pain score | 12 hour postoperative
  Pain score during motion 12 hours postoperatively was assessed using a standard 10 cm linear Visual Analogue Scale, where 0 represents the minimum score and 10 the maximum, with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
VAS Pain score | 24 hour postoperative
  VAS Pain score at rest and motion at immediate, 1, 6, 12, 24 hour postoperatively was assessed using a standard 10 cm linear Visual Analogue Scale, where 0 represents the minimum score and 10 the maximum, with higher scores indicating worse outcomes.
Time to first rescue analgesia | 24 hour postoperative
  The time from the intrathecal injection to the first analgesic intervention
Total analgesics consumption | 24 hour postoperative
  Total analgesics consumption in 24 hour postoperative
Nausea and vomiting incidence | 24 hour postoperative
  Incidence of adverse effect
Pruritus incidence | 24 hour postoperative
  Incidence of adverse effect
Sedation score(Ramsay sedation scale) | 24 hour postoperative
  Sedation was assessed using the Ramsay Sedation Scale, which grades sedation on a scale from 1 to 6 based on the patient's responsiveness to stimuli, higher scores generally indicate deeper sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Piyatida Pirasut, MD, Principal Investigator — Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No